CLINICAL TRIAL: NCT02437734
Title: Virtual Coronary Physiology: an Angiogram is All You Need
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STH16467
Record Dates: First submitted 2015-04-30; First posted 2015-05-08 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Coronary angiography (Other): Selected patients will be asked to undergo Coronary angiography with cardiac magnetic resonance imaging before and after Percutaneous Coronary Intervention. Clinical data collection will happen over a 30 month period.
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — A phase II, observational, analytical study of coronary angiography and computational fluid dynamics in 100 adults with coronary artery disease undergoing coronary angiography.

SUMMARY:
Disease in coronary arteries kills more people in the UK than any other cause. The investigators have developed a computer system ('VIRTU') which predicts blood pressure changes inside coronary arteries. This is important because;

* Doctors make better decisions regarding when and how to treat patients with coronary artery disease if they have these blood pressure measurements
* Currently, Doctors have to insert a metal wire inside the heart to measure artery pressures which is time-consuming and requires special equipment, staff, training and medicines.

Although this invasive technique saves lives and money, more than 95% of patients do not receive the procedure or the benefits it provides.

VIRTU provides a solution to this problem since it only needs X-ray pictures and does not require any wires, drugs, or additional time, equipment or staff. VIRTU has been tested and works but needs improving before it can be used in all patients.

GOALS:

Following, and compared with, our pilot project ((Modelling the significance of coronary artery disease, STH 15740) to:

1. Improve VIRTU's accuracy.
2. Improve VIRTU's speed.
3. Test VIRTU in patients with more complicated coronary disease.

One hundred patients will be recruited from angiography waiting lists and consented before attending for their angiography. The patients will be asked whether their angiogram pictures and pressure measurements maybe used as part of the data collection for this study. The data will be used to validate and develop VIRTU to make it 'patient-ready'. VIRTU will deliver all the advantages of the current invasive technique (i.e. reduced deaths, heart attacks and cost) but, is less invasive and usable in 100% patients.

DETAILED DESCRIPTION:
1. Plan of Investigation Several interacting workstreams will proceed in parallel in this observational, analytical, 36-month study between the University of Sheffield (UoS), Sheffield Teaching Hospitals NHS Foundation Trust (STH), and our collaborators at King's College London (KCL).

   This protocol document outlines the methodology for clinical data collection from patients attending STH. These (fully anonymised) clinical data will then be used to validate and optimise the use of VIRTU by improving its accuracy and speed as well as developing a user-friendly interface. The development work will take place within the UoS and KCL, with no impact on NHS patient, staff or premises after the clinical data collection described below (these subsequent workstreams are detailed in Appendix 1).
2. Study design A phase II, observational, analytical study of coronary angiography and computational fluid dynamics in 100 adults with coronary artery disease undergoing coronary angiography.
3. Methodology (Workstream 1) Clinical data will be collected from the Cardiac Catheter Laboratory (CCL) at STH in a similar manner to which was performed in a pilot project. Therefore, the feasibility of recruitment targets and modelling techniques to be used in this study have already been demonstrated. In this current study, 100 patients with stable CAD of any pattern/severity, potentially suitable for PCI, will be recruited.

   Potential participants will be identified by a member of the care team from pre-admission clinic lists in the cardiac catheter laboratory at the time of diagnostic angiography or referral from another Cardiologist. These patients will be sent a patient information sheet. If they are interested in finding out more about the study, the patients will meet with the Research Nurse or Doctor to discuss the project in more detail and ask questions. At the pre-admission clinic the Research Nurse or Doctor will take informed consent from those patients willing to participate and complete the study recruitment log and the Clinical Details section of the Data Collection Form.

   The patients will then attend for their scheduled PCI at the Northern General Hospital at a later date (usually 2 -3 weeks after the pre-admission clinic). Details of the clinical procedure are below. During the PCI a member of the research team (Dr Gunn, Dr Morton, Dr Morris or Research Nurse) will record the arterial diagrams and procedure details on the second part of the anonymised Data Collection Form.
4. Clinical Procedure Selected patients will be asked to undergo cardiac magnetic resonance imaging before and after PCI, using a standardised protocol. All clinical and angiographic techniques are in routine NHS clinical practice. No experimental techniques will be used. Pre- and post procedure care will not alter from routine elective PCI care.

   The PCI will proceed as normal where indicated, using best contemporary practice, including premedication. The study methods are in routine use for many patients undergoing PCI; and include rotational coronary angiography and pressure wire deployment to assess the physiological significance of lesions. This study merely requires that they be used systematically using standardised methodology.

   Rotational coronary angiography will be recorded in standard single axis rotations (cranial and caudal for left coronary; plane PA for right coronary). An intravenous bolus of 200mcg GTN will be given prior to each run. They will be done on a breath hold, with a rapid hand injection of 10-20mL of contrast. Also, standard, single plane, orthogonal, carefully selected, angiograms will be recorded to guide the procedure. These will be performed at baseline and after stent deployment.

   All major epicardial diseased vessels will be interrogated with a pressure wire (Volcano Corporation). An infusion of adenosine (140mcg/kg/min) will be set up and attached to the intravenous cannula in the hand/arm. The pressure wire will be calibrated against the guide catheter pressure, with the introducing needle removed. The wire will then be advanced across the lesion(s). A bolus of 200mcg GTN will be given and then the iv adenosine infusion started (repeated as necessary since adenosine has very short half life). When the pressures have stabilised, the baseline pressure and flow velocity will be recorded as the wire is withdrawn, while imaging, at 1cm/sec.

   Stent implantation will proceed according to the clinical judgment of the operator, using both the angiographic appearance and the pressure gradient (Fractional Flow Reserve) across any lesions of interest as arbiters. Standard criteria will be used; namely a stenosis that appears to be >50% diameter stenosis in 2 orthogonal projections by eye (or >70% in one) and/or an FFR <0.80. The choice of stent will be at the discretion of the operator.

   After stent deployment, the rotational angiograms and pressure wire pullback will be repeated, using the methods described above. In the case of multi-vessel disease, the pullback will be repeated for the 2nd and the 3rd vessels.
5. Setting for the project Clinical data collection will happen over a 30 month period within Sheffield Teaching Hospitals NHS Foundation Trust, Northern General Hospital. Cardiac Catheter Laboratory will be used for all procedures, because it possesses single axis rotational angiography.
6. Patient population One hundred patients will be recruited from PCI waiting lists.

ELIGIBILITY:
Inclusion Criteria:

* Stable symptoms of coronary ischemia
* Coronary angiographic findings of significant or borderline coronary lesions of any morphology
* Potentially suitable for PCI

Exclusion Criteria:

* Critical ischemia
* Significant valvular heart disease
* Bleeding diathesis
* Terminal cancer
* Pregnancy 6. Lack of informed consent
* Chronic total occlusion of target vessel
* Acute presentation in the previous 60 days
* Intolerance of adenosine, nitrate, iodine based contrast media
* Inability to take dual antiplatelet therapy
* Target vein graft.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2013-08-13 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Intracoronary blood pressures | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nana Theodorou, Study Chair — STH
Locations (1):
- Northern General Hospital, Sheffield, South Yorkshire, United Kingdom